CLINICAL TRIAL: NCT04813588
Title: Comparison of Pantomiming and Easy Onset Treatment on Blocking in Stammering
Brief Title: Comparison of Pantomiming and Easy Onset Treatment
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Riphah International University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: REC/00897 Saba Imtiaz
Record Dates: First submitted 2021-02-16; First posted 2021-03-24 (Actual); Last update posted 2021-03-24 (Actual); Status verified 2021-03

CONDITIONS: Stammering
Keywords: Pantomiming; Easy onset method; Blocking
MeSH Terms: conditions — Stuttering

STUDY DESIGN:
Intervention Model Description: RCT
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Pantomimng (Experimental): In experimental group pantomiming treatment will be administered
  Interventions: Other: Pantomiming
- Easy onset (Active Comparator): In active comparator group easy onset method will be administered
  Interventions: Other: Easy onset

INTERVENTIONS:
Other: Pantomiming — Pantomiming with fluency shaping techniques
  Arms: Pantomimng
Other: Easy onset — Easy onset method with breathing exercises
  Arms: Easy onset

SUMMARY:
This research will give in-depth understanding of pantomiming and easy onset method as an intervention of stuttering and especially blocking. And by comparing both methods, It will also determine that which method is more effective. This research will also improve the overall awareness regarding stuttering

DETAILED DESCRIPTION:
Research participants will be divided into two groups through randomization, Group A & Group B. Base line assessment will be conducted. Intervention will be provided (thrice a week on alternative days).post assessment will be taken and data will be analyzed through SPSS.

ELIGIBILITY:
Inclusion Criteria:

* Participants falling in this category would be added into the study.
* School aged children and adolescents ages between 6 to 18 years(both genders) who stutter with blocking symptoms
* Participant who will be at moderate level of stammering will be included

Exclusion Criteria:

* Participant failing to fall in this category would be excluded of the study.
* Participants with any other medical condition will be excluded

Ages: 6 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 20 (Estimated)
Dates: Start 2021-03-01 (Actual); Primary Completion 2021-05-01 (Estimated); Study Completion 2021-06-01 (Estimated)

PRIMARY OUTCOMES:
The real time analysis | 12 weeks
  Changes from base line "The Real time analysis will use. It will use to assessed the changes in frequency ,duration types and severity of disfluencies in spontaneous speech.The total number of dysfluencies will be divided by the total number of syllables then multiply answer by 100 .Results between 2% showed normal range,8-15% will consider Moderate level, 12% will consider as severe level

CONTACTS AND LOCATIONS:
Overall Officials: Maryam Kiyani, MS/SLP, Principal Investigator — Riphah International University
Locations (1):
- Maryam Nadir Kiyani, Rawalpindi, Punjab Province, Pakistan

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Belyk M, Kraft SJ, Brown S. Stuttering as a trait or state - an ALE meta-analysis of neuroimaging studies. Eur J Neurosci. 2015 Jan;41(2):275-84. doi: 10.1111/ejn.12765. Epub 2014 Oct 28. PMID 25350867
- [Background] 2. Mundada M, Gawali B, Kayte S. Recognition and classification of speech and its related fluency disorders. International Journal of Computer Science and Information Technologies (IJCSIT). 2014;5(5):6764-7.
- [Background] 3. Hudock D, Altieri N, Sun L, Bowers A, Keil C, Kalinowski J. The effect of single syllable silent reading and pantomime speech in varied syllable positions on stuttering frequency throughout utterance productions. Speech Communication. 2015 Dec 1;75:76-83.
- [Background] 4. Waghmare SD, Deshmukh RR, Shrishrimal PP, Waghmare VB, Janvale GB, Sonawane B. A Comparative Study of Recognition Technique Used for Development of Automatic Stuttered Speech Dysfluency Recognition System. Indian Journal of Science and Technology. 2017 Jul;10(21):1-4.
- [Background] Euler HA, Lange BP, Schroeder S, Neumann K. The effectiveness of stuttering treatments in Germany. J Fluency Disord. 2014 Mar;39:1-11. doi: 10.1016/j.jfludis.2014.01.002. Epub 2014 Jan 27. PMID 24759189
- [Background] 6. Kordell J. Outcomes of a Combined Mindfulness, Stuttering Modification, and Fluency Shaping Intervention for Children Who Stutter
- [Background] 7. Keil CM, Hudock D, Altieri N, Seikel AT. The Effects of Pantomine Speech & Silent Reading in Varied Syllable Positions Throughout a Phrase on Stuttering
- [Background] 8. Rifaie NA, Saber AS, El-Din ST, Sallam YA, Algamal AM. Efficacy of the Arabic Modified Fluency Shaping Program in the treatment of stuttering. The Egyptian Journal of Otolaryngology. 2016 Oct 1;32(4):306.
- [Background] 9. Franklin CM. The Effect of Easy Onset Time Treatment on Voice Onset Time in Stuttering.